CLINICAL TRIAL: NCT04566341
Title: Study of Gastrointestinal Dysfunction and Enteric Neural Pathology in Patients With Parkinson's Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Guillermo J. Tearney, MD, PhD, FACC, FCAP, FNAI, Massachusetts General Hospital
Other Study IDs: 2018P001226
Record Dates: First submitted 2020-08-11; First posted 2020-09-28 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Parkinson
Keywords: OCT; Optical Coherence Tomography; TCE; Tethered Capsule Endomicroscopy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Feasibility of OCT TCE in identifying signs of PD: Participants that fulfill our Inclusion/Exclusion criteria will be asked to swallow our Capsule Imaging device.
  Interventions: Device: OCT - TCE

INTERVENTIONS:
Device: OCT - TCE — Participants will be asked to swallow the TCE. They may use mild numbing spray, and lubrication spray to help swallowing. Imaging will be conducted once the TCE is past the pharynx. We will advance the TCE until the stomach and then slowly pull the TCE back up the esophagus. This may be repeated twice.

SUMMARY:
The goal of this research is to determine (1) the feasibility of tethered capsule OCT esophageal imaging in the Parkinson's Disease population; (2) the morphologic changes in the enteric nervous system of the esophagus in patients with Parkinson's disease.

DETAILED DESCRIPTION:
The purpose of this study is to establish the esophageal pathology findings as imaged with tethered capsule microscopy in participants with Parkinson Disease. Images from participants with Parkinson disease will be compared to our previously obtained images in healthy participants to establish the spectrum of esophageal pathologies occurring in participants with Parkinson disease by OCT imaging.

In the case of imaging internal luminal organs, like the esophagus, OCT light is delivered via a long catheter. We have developed a new technique termed Tethered Capsule Endomicroscopy (TCE). TCE involves swallowing a tethered capsule that acquires cross-sectional microscopic images of the entire esophagus as it traverses the luminal organ via peristalsis or is pulled up towards the mouth using tether. The catheter is connected to the imaging system, and the side-viewing optical beam rotates either proximally by a motorized rotary joint or distally by a micro-motor, effectuating circular scanning of the lumen wall. Three-dimensional OCT of the entire length of the lumen can be acquired by simultaneous rotation and translation of the focused OCT beam creating a helical pattern.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease as defined by the United Kingdom PD Society Brain Bank Criteria
* Parkinson Disease Hoehn and Yahr stage 2-4
* Participants on stable dose of Parkinson Disease medications for at least 4 weeks prior to the study screening
* Participants between 40 and 85 years old
* Participants who are capable of giving informed consent

Exclusion Criteria:

* Atypical or secondary Parkinson Disease
* Esophageal fistula and/or esophageal strictures with a luminal stricture diameter that is smaller than the diameter of the capsule
* Recent intestinal resection (within the last six months)
* Prior gastric, esophageal or oropharyngeal surgery
* Inability to swallow capsules
* Pregnancy, according to participant information

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the treating neurologist (a co-investigator) at MGH.
  In addition, an online advertisement seeking volunteers will be listed on rally.partners.org
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of OCT TCE to identify Parkinson's Disease based on image adequacy | Imaging data is collected during the procedure and analyzed within 1 year of collection.
  The image adequacy will be assessed qualitatively (resolution, contrast, etc).
Feasibility of OCT TCE to identify Parkinson's Disease based on morphological changes compared to matched controls | Imaging data is collected during the procedure and analyzed within 1 year of collection.
  The PI will confirm morphologic changes in the enteric nervous system of the esophagus of Parkinson's Disease subjects compared to matched controls. This is a comparison performed by the PI against historical controls, as this imaging technique is too novel to have standard quality grading.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No